CLINICAL TRIAL: NCT03626688
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Ralinepag When Added to PAH Standard of Care or PAH Specific Background Therapy in Subjects With WHO Group 1 PAH
Brief Title: A Study Evaluating the Efficacy and Safety of Ralinepag to Improve Treatment Outcomes in PAH Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ROR-PH-301; APD811-301 (Other: Arena Pharmaceuticals)
Record Dates: First submitted 2018-07-27; First posted 2018-08-13 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: PAH; Pulmonary Hypertension; Pulmonary Arterial Hypertension; Hypertension; Connective Tissue Diseases; Familial Primary Pulmonary Hypertension; Vascular Diseases; Cardiovascular Diseases; Hypertension, Pulmonary; Lung Diseases; Respiratory Tract Disease
Keywords: Prostacyclin; Connective Tissue Disease-Associated; 6 Minute Walk Test; 6 Minute Walk Distance; Pulmonary Vascular Resistance; Right Ventricular Function
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension; Hypertension; Connective Tissue Diseases; Familial Primary Pulmonary Hypertension; Vascular Diseases; Cardiovascular Diseases; Lung Diseases; Respiratory Tract Diseases | interventions — ralinepag

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ralinepag (Experimental): Ralinepag once daily extended-release tablets (oral) 50, 250, and 400 mcg titrated to the highest tolerated dose.
  Interventions: Drug: Ralinepag
- Placebo (Placebo Comparator): Matching placebo tablets (oral)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ralinepag — Active
  Other Names: APD811
  Arms: Ralinepag
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Study ROR-PH-301, ADVANCE OUTCOMES, is designed to assess the efficacy and safety of ralinepag when added to pulmonary arterial hypertension (PAH) standard of care or PAH-specific background therapy in subjects with World Health Organization (WHO) Group 1 PAH.

DETAILED DESCRIPTION:
Study ROR-PH-301 is a multicenter, randomized, double-blind, placebo-controlled study. Subjects who meet entry criteria will be randomly allocated 1:1 to receive ralinepag or placebo, in addition to their standard of care or PAH-specific background therapy, as applicable. The primary endpoint is the time (in days) from randomization to the first adjudicated protocol-defined clinical worsening event. All primary endpoint events will be adjudicated by an independent Clinical Event Committee (CEC) in a blinded fashion. Subjects who have a confirmed primary endpoint event adjudicated by the CEC at any time during the study and all subjects on treatment at the conclusion of the study who have completed the Week 28 Visit (after the target number of confirmed events is achieved) will have the option to enroll in an open-label extension (OLE) study. Subjects who do not choose to participate in the OLE study will discontinue study drug and should remain in the study for long-term follow-up of survival status and will receive standard of care PAH treatment, at the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Evidence of a personally signed and dated informed consent form indicating that the subject has been informed of all pertinent aspects of the study prior to initiation of any study-related procedures.
3. Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures
4. Primary diagnosis of symptomatic PAH.
5. Has had a right heart catheterization (RHC) performed at or within 3 years prior to Screening (RHC will be performed during Screening if not available) that is consistent with the diagnosis of PAH.
6. Has WHO/ NYHA functional class II to IV symptoms.
7. If on PAH-specific background oral therapy, subject is on stable therapy with either an endothelin receptor antagonist (ERA) and/or a phosphodiesterase type 5 inhibitor (PDE5-I) or a soluble guanylate cyclase (sGC) stimulator.
8. Has a 6MWD of ≥150 meters.
9. If taking concomitant medications that may affect the clinical manifestations of PAH (eg, calcium channel blockers, diuretics, digoxin, or L arginine supplementation, beta blockers, angiotensin-converting enzyme inhibitors, or angiotensin II receptor blockers), must be on a stable dose for at least 30 days prior to the Baseline Visit and the dosage maintained throughout the study. The exception is that the dose of diuretics must be stable for at least the 10 days prior to Baseline.
10. Both male and female subjects agree to use a highly effective method of birth control throughout the entire study period from informed consent through to the 30-Day Follow-up Visit, if the possibility of conception exists. Eligible male and female subjects must also agree not to participate in a conception process during the study and for 30 days after the last dose of IMP. Eligible male subjects must agree not to participate in sperm donation for 90 days after the last dose of IMP.

Exclusion Criteria:

1. For subjects with known HIV-associated PAH, a cluster designation 4 (CD4+) T-cell count <200/mm3 within 90 days of Baseline.
2. Must not have 3 or more left ventricular dysfunction risk factors as defined in the study protocol.
3. Has evidence of more than mild lung disease on pulmonary function tests performed within 180 days prior to, or during Screening.
4. Has evidence of thromboembolic disease as determined by a V/Q lung scan or local standard of care diagnostic evaluation at or after diagnosis of PAH.
5. Current diagnosis of ongoing and clinically significant sleep apnea as defined by the Investigator.
6. Male subjects with a corrected QT interval using Fridericia's formula (QTcF) >450 msec and female subjects with a QTcF >470 msec on ECG recorded at Screening and analyzed by the central ECG laboratory. Subjects with evidence of intraventricular conduction delay, defined as a QRS interval greater than 110 msec, will be excluded if the QTcF is >500 msec for both males and females.
7. Severe chronic liver disease (ie, Child-Pugh Class C), portal hypertension, cirrhosis or complications of cirrhosis/portal hypertension (eg, history of variceal hemorrhage, encephalopathy).
8. Confirmed active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV).
9. Subjects with alanine aminotransferase or aspartate aminotransferase ≥3 times the upper limit of normal (ULN) or total bilirubin ≥2 × ULN at Screening.
10. Chronic renal insufficiency as defined by serum creatinine >2.5 mg/dL or requiring dialysis at Screening.
11. Hemoglobin concentration <9 g/dL at Screening.
12. Subjects treated with an IV or SC prostacyclin pathway agent (eg, epoprostenol, treprostinil, or iloprost) or activin signaling inhibitor for PAH at any time prior to Baseline (use in vasoreactive testing is permitted).
13. Subjects currently on or who were treated with an inhaled or oral prostacyclin pathway agent (iloprost, treprostinil, beraprost, or selexipag) for >6 months or within 90 days prior to Baseline.
14. Subject has pulmonary veno-occlusive disease.
15. Malignancy diagnosed and/or treated within 5 years prior to Screening, with the exception of localized non-metastatic basal cell or squamous cell carcinoma of the skin or in-situ carcinoma of the cervix excised with curative intent.
16. Subject tests positive for amphetamine, cocaine, methamphetamine, methylenedioxymethamphetamine or phencyclidine in urine drug screen performed at Screening, or has a recent history (6 months) of alcohol or drug abuse. A subject will not be excluded due to a positive drug screen caused by prescribed medications.
17. Initiation or discontinuation of a cardio-pulmonary rehabilitation program based upon exercise within 90 days prior to Screening and/or planned during study participation.
18. Prior participation in any study of ralinepag or participation in another interventional clinical study with medicinal products within 30 days prior to Screening. Concurrent participation in registry or observational studies is allowed, as long as the subject can fulfill all other entry criteria and comply with all study procedures.
19. Any reason that, in the opinion of the Investigator or Medical Monitor, precludes the subject from participating in the study (eg, any previous or intercurrent medical condition) that may increase the risk associated with study participation or that would confound study analysis or impair study participation or cooperation.
20. Known hypersensitivity to ralinepag or any of the excipients.
21. Life expectancy <12 months based on the Investigator's opinion.
22. Women who are pregnant, lactating or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 728 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Time from randomization to the first adjudicated protocol-defined clinical worsening event | The study duration was event-based. This parameter was assessed from randomization until the conclusion of the study, up to 3 years
  Clinical worsening events are defined as death, nonelective hospital admission for worsening PAH (further defined in clinical study protocol), initiation of parenteral or inhaled prostacyclin pathway agent for treatment of worsening PAH, disease progression (further defined in clinical study protocol), or unsatisfactory long-term clinical response (further defined in clinical study protocol).

SECONDARY OUTCOMES:
Change from Baseline in N-terminal pro-brain natriuretic peptide (NT-proBNP) | Baseline to Week 28
  NT-proBNP was measured at Baseline (prior to starting study drug) and Week 4, 8, 12, and 16, then every 12 weeks thereafter including the End of Study/Early Termination Visit.
Change from Baseline in 6-minute walk distance (6MWD) | Baseline to Week 28
  6MWD was measured at Baseline (prior to starting study drug) and Week 4, 8, 12, and 16, then every 12 weeks thereafter including the End of Study/Early Termination Visit.
Change from Baseline in WHO/New York Heart Association (NYHA) Functional Class | Baseline to Week 28
  The severity of PAH was graded according to the functional status of the subject and assessed at every visit.
Shift and proportion of subjects who attain all 3 of the following: NT-proBNP level <300 pg/mL, 6MWD >440 meters, and WHO/NYHA Functional Class I or II | Baseline to Week 28
  Data from NT-proBNP, 6MWD, and WHO/NYHA functional class assessment were compiled as a composite endpoint at visits through Week 28.
Registry to Evaluate Early and Long-term PAH Disease Management (REVEAL) risk score | Baseline to Week 28
  Data from NT-proBNP, 6MWD, WHO/NYHA functional class, systolic blood pressure, heart rate, and estimated glomerular filtration rate values collected at visits through Week 28 were used to calculate the composite REVEAL risk score.
Clinical improvement as defined by the absence of clinical worsening and fulfillment of at least 2 of the 3 of the following: increase in 6MWD ≥10% or ≥30 m, improvement to or maintenance of WHO FC I or II, and decrease in NT-proBNP by at least 30%. | Baseline to Week 28
  Data from 6MWD, WHO/NYHA functional class assessment, and NT-proBNP were compiled as a composite endpoint at visits through Week 28.
Change from Baseline in health-related quality of life as measured by patient-reported outcomes. | Baseline to Week 28
  Quality of life was assessed using patient-reported outcomes at Baseline (prior to starting study drug) and Week 16, then every 12 weeks thereafter including the End of Study/Early Termination Visit.
Time to first all-cause nonelective hospitalization | The study duration was event-based. This parameter was assessed from randomization until the conclusion of the study (when the target number of adjudicated events was achieved, as defined in the study protocol).
  All nonelective hopsitalizations during the study period were collected.
Time to all-cause mortality | The study duration was event-based. This parameter was assessed from randomization until the conclusion of the study (when the target number of adjudicated events was achieved, as defined in the study protocol).
  All deaths during the study period were collected.
Change from Baseline in heart rate recovery (HRR) following completion of the 6MWT | Baseline to Week 28
  HRR was measured at Baseline (prior to starting study drug) and Week 4, 8, 12, and 16, then every 12 weeks thereafter including the End of Study/Early Termination Visit.
Safety and tolerability of ralinepag in subjects with PAH | Baseline to Week 28
  Safety and tolerability were assessed by adverse events.

CONTACTS AND LOCATIONS:
Locations (209):
- United States (68):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - UCSD Health Sciences, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Keck Hospital of USC, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - University of California, Irvine, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - SBPA Research LLC, Santa Barbara, California
  - Stanford Healthcare, Stanford, California
  - LA Biomedical Research Institute Harbor-UCLA Medical Center, Torrance, California
  - University of Colorado Hospital, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Central Florida Pulmonary Group, Orlando, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Piedmont Healthcare Pulmonary and Critical Care Research, Austell, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Ascension Alexian Brothers, Elk Grove Village, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Community Health Network Cancer Center North, Indianapolis, Indiana
  - St. Vincent Medical Group, Inc., Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Kentuckiana Pulmonary Research Center, Louisville, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - Chest Medicine Associates, South Portland, Maine
  - University of Maryland Medical Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - Spectrum Health Medical Group, Grand Rapids, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Medical Center, Omaha, Nebraska
  - University of New Mexico, Albuquerque, New Mexico
  - Winthrop Hospital, Mineola, New York
  - NYU Langone Medical Center, New York, New York
  - Weill-Cornell-New York Presbyterian Hospital, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - University of Rochester, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - University of Cincinnati-Medical Science Building, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Oregon Clinic-Pulmonary West, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Statcare Pulmonary Consultants, Knoxville, Tennessee
  - Ascension Texas Cardiovascular, Austin, Texas
  - Baylor University Medical Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - The Methodist Hospital Research Institute, Houston, Texas
  - Vermont Lung Center, Colchester, Vermont
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia
  - Carilion Clinic Pulmonary and Sleep Medicine, Roanoke, Virginia
  - Medical College of Wisconsin/Froedtert Hospital, Milwaukee, Wisconsin
- Argentina (12):
  - Hospital Italiano, Ciudad Autonoma Buenos Aires, Buenos Aires
  - Instituto de Investigaciones Clinicas Mar del Plata, Mar del Plata, Buenos Aires
  - Sanatorio Parque, Rosario, Santa Fe Province
  - Sanatorio de la Trinidad Mitre, Buenos Aires
  - Cardiologia Palmero, Caba
  - Hospital Britanico de Buenos Aires, Ciudad Autonoma Buenos Aires
  - Fundacion Respirar, Ciudad Autonoma Buenos Aires
  - Fundacion Favaloro, Ciudad Autonoma Buenos Aires
  - Instituto de Cardiologia de Corrientes, Corrientes
  - Hospital Italiano de Cordoba, Córdoba
  - Hospital Privado Centro Medico de Cordoba S.A, Córdoba
  - Hospital PROVINCIAL "Dr. Jose Maria Cullen", Santa Fe
- Australia (11):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Macquarie University, Macquarie, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Austria (3):
  - Medizinische Universität Innsbruck, Innsbruck
  - Ordensklinikum Linz GmbH - Elisabethinen, Fadingerstrasse 1, Linz
  - AKH Wien, Innere Med. II, Kardiologie, Währingergürtel 18-20, Vienna
- Belgium (2):
  - Cliniques Universitaires de Bruxelles Hopital Erasme, Brussels
  - UZ Leuven, UZ Leuven Campus Gasthuisberg, Herestraat 49, Leuven
- Brazil (7):
  - HC-UFG - Hospital das Clínicas da Universidade Federal de Goiás, Goiânia, Goiás
  - Instituto das Pequenas Missionárias de Maria Imaculada - Hospital Madre Teresa, Belo Horizonte, Minas Gerais
  - Hospital Sao Lucas da PUC-RS, Porto Alegre, R.S
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - UNESP-Faculdade de Medicina da Universidade Estadual Paulista Campus Botucatu, Botucatu, São Paulo
  - Hospital Sao Paulo, São Paulo, São Paulo
  - Instituto do Coracao, São Paulo, São Paulo
- Bulgaria (2):
  - MHAT - "National Heart Hospital" EAD, 65, Konyovitza Str., Sofia
  - MHAT "Sveta Anna" Sofia AD, Sofia
- Canada (5):
  - Peter Lougheed Centre, Calgary, Alberta
  - LHSC - Victoria Hospital, London, Ontario
  - University Health Network-Toronto General Hospital, Toronto, Ontario
  - SMBD Jewish General Hospital d/b/a Jewish General Hospital, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec, Québec, Quebec
- Instiuto Nacional del Torax, Providencia, Santiago de Chile, Chile
- China (5):
  - Beijing Shijitan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing
- Croatia (2):
  - Clinical Hospital Dubrava Zagreb, Avenija G.Šuška 6, Zagreb
  - University Clinic for Pulmonary Diseases, Jordanovac 104, Zagreb
- Vseobecna fakultni nemocnice v Praze, II. interni klinika kardiologie a angiologie VFN a 1. LF UK, U nemocnice 2, Prague, Czechia
- Denmark (2):
  - Århus Universitetshospital, Aarhus
  - Copenhagen University Hospital (Rigshospitalet), Copenhagen
- France (11):
  - CHU de Strasbourg - Nouvel Hôpital Civil, Ctre de competence Hypertension Arterielle Pulmona, 1 place de l Hopital, Strasbourg, Bas Rhin
  - CHU de Grenoble - Hôpital Albert Michallon, Clinique de Cardiologie, Boulevrad de la Chantourne, Grenoble, Isere
  - CHU Nancy - Hôpital de Brabois Adultes, Pneumologie- Oncologie Médicale, Rue du Morvan, Vandœuvre-lès-Nancy, Meurthe Et Moselle
  - CHU de Saint-Etienne - Hopital Nord, Service de Medecine vasculaire et therapeutique, 81 Avenue A. Raimond, Saint-Étienne-de-Montluc, Pays de la Loire Region
  - CHU Lyon - Hôpital Cardio-Vasculaire et Pneumologique Louis Pradel, Service de Pneumologie, 59 Boulevard Pinel, Bron, Rhone
  - CHU de Rouen - Hôpital Charles Nicolle, Rouen, Seine Maritime
  - Groupement Hospitalier Sud - Hôpital Bicêtre, Le Kremlin-Bicêtre, Val De Marne
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - CHU de Brest - Hôpital de la Cavale Blanche, Brest
  - CHRU de Lille - Hopital Cardiologique, Lille
  - Hôpital Nord - CHU Marseille, Marseille
- Germany (8):
  - Thoraxklinik-Heidelberg Zentrum für Pulmonale Hypertonie, Heidelberg, Baden-Wurttemberg
  - Universitätsmedizin Greifswald, Greifswald, Mecklenburg-Vorpommern
  - Universitaetsmedizin der Johannes-Gutenberg-Universitaet Mainz, Zentrum für Kardiologie I, Centrum für Thrombose und Hämostase (CTH), Langenbeckstrasse 1, Mainz, Rhineland-Palatinate
  - Universitaetsklinikum des Saarlandes, Innere Medizin V, IMED, Kirrberger Strasse 100, Gebäude 41, Homburg, Saarland
  - Universitätsklinikum Leipzig, Medizinische Klinik II, Pneumologie, Leipzig, Saxony
  - Schwarzwald-Baar Klinikum, Donaueschingen
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
- Greece (4):
  - "Onasseio" Cardiosurgery Hospital, Hemodynamic Research and Interventional Cardiology Dept., 356, Syggrou Avenue, Athens, Kallithea
  - University General Hospital of Alexandroupolis, Alexandroupoli
  - University General Hospital Attikon, Chaïdári
  - AHEPA General Hospital of Thessaloniki, A' Cardiology Clinic, 1 St. Kyriakidi Street, Thessaloniki
- Hungary (3):
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ Családorvosi Intézet és Rendelő, Szeged, Csongrád-Csanád
  - Gottsegen György Országos Kardiovaszkuláris Intézet, Budapest
  - Pecsi Tudomanyegyetem, Szivgyogyaszati Klinika, Ifjusag u. 13., Pécs
- Israel (5):
  - The Lady Davis Carmel Medical Center, 7 Michal st., Haifa
  - Hadassah Ein Kerem Medical Center, Kiryat Hadassah, Jerusalem
  - Meir Medical Center, 59 Tshernichovski st., Kfar Saba
  - Rabin Medical Center-Beilinson Campus, Pulmonary Institute, 39 Jabotinsky St Ground floor, Petah Tikva
  - Tel Aviv Sourasky Medical Center, 6 Weizmann St., Tel Aviv
- Italy (7):
  - Istituto Mediterraneo Trapianti e Terapie a Alta Specializzazione (IRCCS-ISMETT), Palermo, PA
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Foggia, S.C. di Cardiologia, Viale Luigi Pinto, 1, Foggia
  - IRCC Ospedale Policlinico San Martino, Genova
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Via Francesco Sforza 35, Milan
  - Azienda Socio Sanitaria Territoriale di Monza (Presidio San Gerardo), Monza
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliera Universitaria Policlinico Umberto I - Università di Roma La Sapienza, Viale del Policlinico, 155, Roma
- Mexico (4):
  - CICUM San Miguel, Guadalajara, Jalisco
  - Instituto Nacional de Cardiologia Dr Ignacio Chavez Rivera, Mexico City, Mexico City
  - Instituto Nacional de Ciencias Médicas y Nutricion Dr. Salvador Zubiran, Mexico City, Mexico City
  - Unidad de Investigacion Clinica en Medicina, S.C., Monterrey, N.L.
- VU Medisch Centrum, De Boelelaan 1117, Amsterdam, Netherlands
- Poland (5):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Klinika Kardiologii z Oddzialem Intensywnego Nazdoru Kardiologicznego, M. Sklodowskiej 24a, Bialystok
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II, Oddział Kliniczny Chorób Serca i Naczyń z Pododdziałem Intensywnego Nadzoru Kardiologicznego, Pradnicka 80, Krakow
  - NZOZ Europejskie Centrum Zdrowia, ul. Borowa 14/18, Otwock
  - Szpital Kliniczny Przemienienia Panskiego Uniwersytetu Medycznego im. Karola Marcinkowskiego w Poznaniu, Oddzial Kardiologii - F, ul. Dluga 1/2, Poznan
  - Premium Clinic Wrocław CM, Podwale 83/17, Wroclaw
- Portugal (4):
  - Hospital Garcia de Orta, E.P.E, Almada
  - Centro Hospitalar e Universitário de Coimbra, E.P.E., Coimbra
  - Centro Hospitalar Universitário Lisboa Norte, E.P.E. Hospital Pulido Valente, Lisbon
  - Centro Hospitalar de Santo António E.P.E., Porto
- Romania (4):
  - Institutul de Urgenta pentru Boli Cardiovasculare "Prof. Dr. C.C. Iliescu", Sos. Fundeni nr. 258, Bucharest
  - Institutul de Pneumoftiziologie "Marius Nasta", Sos. Viilor nr. 90, Sector 5, Bucharest
  - Institutul Inimii "Niculae Stancioiu" Cluj-Napoca, Cardiologie, Str. Motilor nr. 19-21, Cluj-Napoca
  - Spitalul Clinic de Boli Infectioase si Pneumoftiziologie "Dr. Victor Babes" Timisoara, Str. Gheorghe Adam nr. 13, Timișoara
- Serbia (3):
  - Clinical Center of Serbia, Koste Todorovica 8, Belgrade
  - Clinical Center Zemun. Clinic for internal medicine, Department of Cardiology, Belgrade
  - Institute for Pulmonary Diseases of Vojvodina, Put Dr Goldmana 4, Kamenitz
- Singapore (2):
  - National University Hospital, Singapore
  - National Heart Centre, Singapore
- South Korea (3):
  - Samsung Medical Center, Seoul, Gangnam-gu
  - Seoul National University Hospital, Seoul, Jongno-gu
  - Gachon University Hospital Gil Medical Center, Incheon, Namdong-gu
- Spain (4):
  - Hospital Universitari Vall d'Hebron, Respiratory Dept., Passeig Vall d'Hebron,119-129, Neumologia, Barcelona
  - Hospital Clinic de Barcelona, C/ Villarroel, 170, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospoital Universitari i Politecnic La Fe, Valencia
- Sweden (3):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Linköping Universitetssjukhuset, Linköping
  - Norrlands Universitetssjukhus, Hjärtcentrum, Umeå
- Taiwan (2):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- Turkey (Türkiye) (7):
  - Osmangazi Uni Medical Faculty, Eskişehir, Odunpazari
  - Balcalı, Çukurova Üniversitesi Kardiyoloji ABD, Adana, Saricam
  - Mersin Üniversitesi Tip Fakültesi Ciftlikköy Kampüsü, Mersin, Yenisehir
  - Gazi University Medical Faculty Hospital, Ankara
  - Uludag Universitesi Tip Fakültesi, Gorukle Kampusu, Bursa
  - Marmara Universitesi Istanbul Pendik Egitim ve Arastirma Hastanesi, Istanbul
  - Dokuz Eylul Universitesi Tip Fakultesi, Mithatpasa caddesi Inciralti Balcova, Izmir
- Ukraine (3):
  - CE Dniprop RCC&C Center of Dniprop RC Dept of Card SI DMA of MOHU, Chair of Internal Medicine 3, 28, Knyazya Volodymyra Velykogo St., Dnipro
  - SI F.H.Yanovskyi National Institute of Phthisiology and Pulmonology of NAMSU, Clinical and Functional Dept, 10, Amosova St., Kyiv
  - Communal Noncommercial Enterprise of Lviv Regional Council Lviv Clinical Hospital, Dept of Cardiology, D.Halytskyi Lviv NMU, Ch of Internal Medicine #1, 7, Chernihivska str., Lviv
- United Kingdom (5):
  - Royal Free London NHS Foundation Trust, Pond Street, London, Greater London
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Sir William Leech Lung Research Centre, Newcastle upon Tyne, Tyne and Wear
  - Golden Jubilee National Hospital, Glasgow, West Dunbartonshire
  - Royal Brompton Hospital, London
  - Imperial College Healthcare NHS Trust, London